CLINICAL TRIAL: NCT05080894
Title: Early Domestic Rehabilitation Using Virtual Reality for Patients With Anterior Cruciate Ligament Reconstruction: a Randomized Controlled Trial
Brief Title: Virtual Reality Rehabilitation for Patients With Anterior Cruciate Ligament Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut d'Investigacions Biomèdiques August Pi i Sunyer (Other)
Collaborators: Fundación Mutua Madrileña (Other)
Responsible Party: Principal Investigator, Prof. Maria V. Sanchez-Vives, Professor, Institut d'Investigacions Biomèdiques August Pi i Sunyer
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCB-2019-0670
Record Dates: First submitted 2021-09-20; First posted 2021-10-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Knee Injuries
Keywords: virtual reality; embodiment; rehabilitation; anterior cruciate ligament reconstruction
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality (Experimental): Daily 20-minute sessions of virtual reality based rehabilitation for the first 4 weeks post-operatively + standard rehabilitation protocol
  Interventions: Device: Virtual reality
- Standard intervention (No Intervention): Standard rehabilitation protocol only

INTERVENTIONS:
Device: Virtual reality — Embodiment of a healthy virtual body in virtual reality and action observation/motor imagery of the subject's virtual body performing high-level lower limb exercises.
  Arms: Virtual reality

SUMMARY:
The purpose of this study is to ascertain whether 4 weeks of daily virtual-reality-based rehabilitation at home improves disability in the early stages of recovery from anterior cruciate ligament reconstruction surgery compared with standard care.

DETAILED DESCRIPTION:
After being informed about the study and potential risks and benefits, patients giving written informed consent will be randomized to one of two groups in a 1:1 ratio. The treatment group will perform daily a 20-minute rehabilitation session in virtual reality, in which they will observe their virtual body performing a series of exercises they would otherwise be unable to perform in real life. Both groups will also undergo the standard rehabilitation protocol. The investigators will assess for differences between groups in self-reported disability, knee range of motion, and quadriceps strength at baseline, 4 weeks, 12 weeks and 9 months.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-40 (either sex)
* Post-operative anterior cruciate ligament reconstruction (autograft), either bone-patellar tendon-bone graft or semitendinosus (hamstring) graft

Exclusion Criteria:

* Patients with significant cognitive deficit (MEC<24).
* Patients with epilepsy or severe vision problems
* Pregnant patients
* Previous surgery on the reconstructed knee, excluding arthroscopy
* Previous anterior cruciate ligament reconstruction on either knee
* Sustained concurrent injury to the contralateral knee
* Concomitant collateral ligament and/or meniscal repair
* Presence of symptomatic tibiofemoral osteoarthritis

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
The International Knee Documentation Committee (IKDC) Subjective Knee Form | Baseline (day 1 post-surgery)
  Patient-completed tool, which contains sections on knee symptoms/pain, function, and sports activities. Scores range from 0 points (lowest level of function or highest level of symptoms) to 100 points (highest level of function and lowest level of symptoms).
The International Knee Documentation Committee (IKDC) Subjective Knee Form | 4 weeks
  Patient-completed tool, which contains sections on knee symptoms/pain, function, and sports activities. Scores range from 0 points (lowest level of function or highest level of symptoms) to 100 points (highest level of function and lowest level of symptoms).
The International Knee Documentation Committee (IKDC) Subjective Knee Form | 12 weeks
  Patient-completed tool, which contains sections on knee symptoms/pain, function, and sports activities. Scores range from 0 points (lowest level of function or highest level of symptoms) to 100 points (highest level of function and lowest level of symptoms).
The International Knee Documentation Committee (IKDC) Subjective Knee Form | 9 months
  Patient-completed tool, which contains sections on knee symptoms/pain, function, and sports activities. Scores range from 0 points (lowest level of function or highest level of symptoms) to 100 points (highest level of function and lowest level of symptoms).

SECONDARY OUTCOMES:
Isometric quadriceps strength | Baseline
  Measured knee extension strength with a handheld dynamometer, expressed as peak force (Newtons)
Isometric quadriceps strength | 4 weeks
  Measured knee extension strength with a handheld dynamometer, expressed as peak force (Newtons)
Isometric quadriceps strength | 12 weeks
  Measured knee extension strength with a handheld dynamometer, expressed as peak force (Newtons)
Isometric quadriceps strength | 9 months
  Measured knee extension strength with a handheld dynamometer, expressed as peak force (Newtons)
Knee extension active range of motion | Baseline
  Measured with a digital goniometer (smartphone app)
Knee extension active range of motion | 4 weeks
  Measured with a digital goniometer (smartphone app)
Knee extension active range of motion | 12 weeks
  Measured with a digital goniometer (smartphone app)
Knee extension active range of motion | 9 months
  Measured with a digital goniometer (smartphone app)
Time taken to return to sporting activity | 9 months
  Taken retrospectively at 9 months, number of days from surgery to full return to sport
Kinesiophobia | Baseline
  Fear of movement as measured with the Tampa scale of kinesiophobia
Kinesiophobia | 4 weeks
  Fear of movement as measured with the Tampa scale of kinesiophobia
Kinesiophobia | 12 weeks
  Fear of movement as measured with the Tampa scale of kinesiophobia
Kinesiophobia | 9 months
  Fear of movement as measured with the Tampa scale of kinesiophobia

CONTACTS AND LOCATIONS:
Overall Officials: Maria V. Sanchez-Vives, Principal Investigator — Institut d'Investigacions Biomèdiques August Pi i Sunyer
Locations (1):
- IDIBAPS, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No